CLINICAL TRIAL: NCT03515551
Title: A Phase I/II Study of IMCnyeso, HLA- A*0201-Restricted, NY-ESO-1- and LAGE-1A-specific Soluble T Cell Receptor and Anti-CD3 Bispecific Molecule, in HLA-A*0201 Positive Patients With Advanced NY-ESO-1 and/or LAGE - 1A Positive Cancer
Brief Title: Safety and Efficacy of IMCnyeso in Advanced NY-ESO-1 and/or LAGE-1A Positive Cancers
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Strategic decision to stop development and not based on any safety concerns
Sponsor: Immunocore Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IMCnyeso-101
Record Dates: First submitted 2018-04-05; First posted 2018-05-03 (Actual); Results first posted 2022-03-11 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Select Advanced Solid Tumors
Keywords: IMCnyeso; Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1: Dose Escalation (Experimental): Four fixed-dose, dose escalation cohorts (Cohorts 1 to 4) and 3 intrapatient dose escalation cohorts (Cohorts 5 to 7) to establish the MTD/RP2D of IMCnyeso.
  Interventions: Drug: IMCnyeso
- Phase 2: Dose Expansion (Experimental): Three planned cohorts treated at the RP2D to make a preliminary assessment of the anti-tumor activity of IMCnyeso. Phase 2 was not initiated and data were not collected.
  Interventions: Drug: IMCnyeso

INTERVENTIONS:
Drug: IMCnyeso — Weekly IV infusions of IMCnyeso

SUMMARY:
IMCnyeso is a bispecific fusion protein designed for the treatment of cancers that express NY-ESO-1 and/or LAGE-1A. This was a first-in-human trial designed to evaluate the safety and efficacy of IMCnyeso in HLA-A*02:01-positive adult participants whose cancer is positive for NY-ESO-1 and/or LAGE-A1.

DETAILED DESCRIPTION:
This was planned to be a multi-center, open label, dose finding Phase 1/2 study of single agent IMCnyeso administered in participants with NY-ESO-1 and/or LAGE-A1 positive tumors. The primary objective of the dose escalation phase (Phase 1) was to determine the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) of IMCnyeso in participants with advanced solid tumors. Preliminary efficacy was to be evaluated in Phase 2. The study was terminated early (prior to initiation of Phase 2) by the Sponsor as a strategic decision (not based on any safety signal).

ELIGIBILITY:
Inclusion Criteria:

1. HLA-A*0201 positive
2. NY-ESO-1 and/or LAGE-1A positive tumor
3. ECOG PS 0 or 1
4. Selected advanced solid tumors
5. Relapsed from, refractory to, or intolerant of standard therapy
6. If applicable, must agree to use highly effective contraception

Exclusion Criteria:

1. Symptomatic or untreated central nervous system metastasis
2. Inadequate washout from prior anticancer therapy
3. Significant ongoing toxicity from prior anticancer treatment
4. Impaired baseline organ function as evaluated by out-of-range laboratory values
5. Clinically significant cardiac disease
6. Active infection requiring systemic antibiotic therapy
7. Known history of human immunodeficiency virus (HIV)
8. Active hepatitis B virus (HBV) or hepatitis C virus (HCV)
9. Ongoing treatment with systemic steroids or other immunosuppressive therapies
10. Significant secondary malignancy
11. Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2021-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Immunocore Ltd
Locations (12):
- United States (8):
  - University of Colorado Hospital, Aurora, Colorado
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - UPMC - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Tennessee Oncology NASH - SCRI, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada
- United Kingdom (3):
  - Sarah Cannon Research Institute UK, London
  - The Christie Hospital, Manchester
  - Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lopez JS, Milhem M, Butler MO, Thistlethwaite F, Van Tine BA, D'Angelo SP, Johnson ML, Sato T, Arkenau HT, Edukulla R, Wustner J, Marshall S, Rodon J. Phase 1 study of IMCnyeso, a T cell receptor bispecific ImmTAC targeting NY-ESO-1-expressing malignancies. Cell Rep Med. 2025 Apr 15;6(4):101994. doi: 10.1016/j.xcrm.2025.101994. Epub 2025 Mar 6. PMID 40054461

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The sponsor elected to not proceed with the efficacy determining expansion phase (Phase 2) of IMCnyeso-101 for strategic reasons. Phase 2 data were not collected. As of 25 Mar 2021, further enrollment into the Phase 1 dose escalation phase was discontinued and last patient visit was 10 June 2021. Participants who were receiving study drug were allowed to continue treatment until unacceptable toxicity, disease progression, or other reason to discontinue occurred.
Pre-assignment Details: There were a total of 28 unique participants; one participant from the 10 mcg cohort was sequentially enrolled in the 30-100 mcg cohort.
Groups:
- Phase 1: IMCnyeso 3 mcg: Single-agent IMCnyeso at 3 mcg dosed weekly intravenously on Days 1, 8, 15, and 22 of each 4-week cycle using a fixed-dose regimen
- Phase 1: IMCnyeso 10 mcg: Single-agent IMCnyeso at 10 mcg dosed weekly intravenously on Days 1, 8, 15, and 22 of each 4-week cycle using a fixed-dose regimen
- Phase 1: IMCnyeso 30 mcg: Single-agent IMCnyeso at 30 mcg dosed weekly intravenously on Days 1, 8, 15, and 22 of each 4-week cycle using a fixed-dose regimen
- Phase 1: IMCnyeso 100 mcg: Single-agent IMCnyeso at 100 mcg dosed weekly intravenously on Days 1, 8, 15, and 22 of each 4-week cycle using a fixed-dose regimen
- Phase 1: IMCnyeso 30-100 mcg: IMCnyeso administered intravenously on Days 1, 8, 15, and 22 of each 4-week cycle using an intrapatient escalation regimen (30 mcg on Cycle 1 Day 1, then 100 mcg starting on Cycle 1 Day 8)
- Phase 1: IMCnyeso 30-100-180 mcg: IMCnyeso administered intravenously on Days 1, 8, 15, and 22 of each 4-week cycle using an intrapatient escalation regimen (30 mcg on Cycle 1 Day 1, then 100 mcg on Cycle 1 Day 8, then 180 mcg starting on Cycle 1 Day 15)
- Phase 1: IMCnyeso 30-100-300 mcg: IMCnyeso administered intravenously on Days 1, 8, 15, and 22 of each 4-week cycle using an intrapatient escalation regimen (30 mcg on Cycle 1 Day 1, then 100 mcg on Cycle 1 Day 8, then 300 mcg starting on Cycle 1 Day 15)
Period: Overall Study
Arm/Group | Phase 1: IMCnyeso 3 mcg | Phase 1: IMCnyeso 10 mcg | Phase 1: IMCnyeso 30 mcg | Phase 1: IMCnyeso 100 mcg | Phase 1: IMCnyeso 30-100 mcg | Phase 1: IMCnyeso 30-100-180 mcg | Phase 1: IMCnyeso 30-100-300 mcg
Started | 4 | 3 | 5 | 3 | 5 (1 participant from the 10 mcg cohort was sequentially enrolled in the 30-100 mcg cohort and is counted as starting in both columns; reason for study discontinuation recorded as part of 30-100 mcg cohort.) | 4 | 5
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 3 | 5 | 3 | 5 | 4 | 5
Not completed — Death | 4 | 1 | 2 | 2 | 2 | 4 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Study ended by sponsor | 0 | 0 | 2 | 1 | 3 | 0 | 3
Not completed — Sequential enrollment in 30-100 mcg cohort | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set includes all participants assigned to treatment who receive at least 1 full or partial dose of study drug; one participant that sequentially enrolled in two cohorts (10 mcg and 30-100 mcg) is represented in the 30-100 mcg cohort.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1: IMCnyeso 3 mcg | Phase 1: IMCnyeso 10 mcg | Phase 1: IMCnyeso 30 mcg | Phase 1: IMCnyeso 100 mcg | Phase 1: IMCnyeso 30-100 mcg | Phase 1: IMCnyeso 30-100-180 mcg | Phase 1: IMCnyeso 30-100-300 mcg | Total
Number analyzed (Participants) | 4 | 2 | 5 | 3 | 5 | 4 | 5 | 28
Age, Customized [Count of Participants; unit: Participants]
  18-64 years old | 4 | 2 | 5 | 2 | 3 | 3 | 4 | 23
  65-84 years old | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 1 | 2 | 0 | 4 | 12
  Male | 2 | 1 | 3 | 2 | 3 | 4 | 1 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 4 | 2 | 3 | 3 | 5 | 3 | 5 | 25
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 4 | 2 | 5 | 3 | 5 | 4 | 5 | 28
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Original cancer diagnosis [Count of Participants; unit: Participants]
  Melanoma | 0 | 0 | 0 | 1 | 1 | 2 | 3 | 7
  Synovial sarcoma | 4 | 2 | 5 | 2 | 3 | 2 | 2 | 20
  Urothelial carcinoma | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Non-small cell lung cancer | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number of Participants With Dose-limiting Toxicities
Description: Dose-limiting toxicities were defined as an adverse event or abnormal laboratory value assessed as having a suspected relationship to study drug that occurs within the evaluation period, from the first dose up until Day 28 after the first dose
Time Frame: Up to 35 months
Population: The Safety Analysis Set includes all participants who received at least 1 full or partial dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: IMCnyeso 3 mcg | Phase 1: IMCnyeso 10 mcg | Phase 1: IMCnyeso 30 mcg | Phase 1: IMCnyeso 100 mcg | Phase 1: IMCnyeso 30-100 mcg | Phase 1: IMCnyeso 30-100-180 mcg | Phase 1: IMCnyeso 30-100-300 mcg
Number analyzed (Participants) | 4 | 3 | 5 | 3 | 5 | 4 | 5
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 2

2. Primary Outcome: Phase 1: Number of Participants With Adverse Events
Description: Treatment-emergent adverse events are defined as any adverse event (AE) that started after the first dose of study drug up to 30 days after last dose of study drug, including abnormal laboratory values, vital signs, or electrocardiogram results. AE severity is graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03.
Time Frame: Up to 35 months
Population: The Safety Analysis Set includes all participants who received at least 1 full or partial dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: IMCnyeso 3 mcg | Phase 1: IMCnyeso 10 mcg | Phase 1: IMCnyeso 30 mcg | Phase 1: IMCnyeso 100 mcg | Phase 1: IMCnyeso 30-100 mcg | Phase 1: IMCnyeso 30-100-180 mcg | Phase 1: IMCnyeso 30-100-300 mcg
Number analyzed (Participants) | 4 | 3 | 5 | 3 | 5 | 4 | 5
Participants
  Any treatment-emergent adverse event (TEAE) | 4 | 3 | 5 | 3 | 5 | 4 | 5
  Any TEAE Grade ≥3 | 3 | 1 | 1 | 3 | 3 | 4 | 4
  Any TEAE leading to death | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Phase 1: Number of Participants With No Dose Interruptions or Reductions
Description: Tolerability of study treatment was assessed by summarizing the number of participants with no treatment dose interruptions and dose reductions
Time Frame: Up to 35 months
Population: The Safety Analysis Set includes all participants who received at least 1 full or partial dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: IMCnyeso 3 mcg | Phase 1: IMCnyeso 10 mcg | Phase 1: IMCnyeso 30 mcg | Phase 1: IMCnyeso 100 mcg | Phase 1: IMCnyeso 30-100 mcg | Phase 1: IMCnyeso 30-100-180 mcg | Phase 1: IMCnyeso 30-100-300 mcg
Number analyzed (Participants) | 4 | 3 | 5 | 3 | 5 | 4 | 5
Participants
  No dose interruption at any time | 2 | 0 | 0 | 2 | 2 | 0 | 0
  No dose reduction at any time | 4 | 3 | 5 | 3 | 4 | 4 | 3

4. Primary Outcome: Phase 2: Best Overall Response (BOR)
Description: Best overall response per RECIST v.1.1
Time Frame: Up to 35 months
Population: The study was terminated during Phase 1 due to strategic reasons; data were not collected or analyzed for any Phase 2 outcome measures.
Groups:
- Phase 2: Dose Expansion: Three planned cohorts treated at the RP2D to make a preliminary assessment of the anti-tumor activity of IMCnyeso. The Phase 2 arm was not initiated.
Arm/Group | Phase 2: Dose Expansion
Number analyzed (Participants) | 0

5. Secondary Outcome: Phase 2: Number of Participants With Adverse Events
Description: Treatment-emergent adverse events are defined as any adverse event (AE) that started after the first dose of study drug up to 30 days after last dose of study drug, including abnormal laboratory values, vital signs, or electrocardiogram results.
Time Frame: Up to 35 months
Population: as for outcome 4
Arm/Group | Phase 2: Dose Expansion
Number analyzed (Participants) | 0

6. Secondary Outcome: Phase 2: Number of Participants With No Dose Interruptions or Reductions
Description: as for outcome 3
Time Frame: Up to 35 months
Population: as for outcome 4
Arm/Group | Phase 2: Dose Expansion
Number analyzed (Participants) | 0

7. Secondary Outcome: Phase 1: Number of Participants With Best Overall Response (BOR)
Description: Number of participants with best overall response, including complete response, partial response, stable disease, and progressive disease, based on local Investigator assessment as defined in RECIST v.1.1.
Time Frame: Up to 35 months
Population: The Full Analysis Set includes all participants assigned to treatment who receive at least 1 full or partial dose of study drug and for which evaluation was able to be made for at least 1 post-baseline tumor assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: IMCnyeso 3 mcg | Phase 1: IMCnyeso 10 mcg | Phase 1: IMCnyeso 30 mcg | Phase 1: IMCnyeso 100 mcg | Phase 1: IMCnyeso 30-100 mcg | Phase 1: IMCnyeso 30-100-180 mcg | Phase 1: IMCnyeso 30-100-300 mcg
Number analyzed (Participants) | 4 | 3 | 5 | 3 | 5 | 4 | 5
Participants
  Complete Response | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Stable Disease | 0 | 0 | 2 | 0 | 2 | 0 | 1
  Progressive Disease | 3 | 3 | 3 | 3 | 3 | 3 | 3
  Non-evaluable | 1 | 0 | 0 | 0 | 0 | 1 | 1

8. Secondary Outcome: Phase 1 and Phase 2: Progression-free Survival
Description: Progression-free survival is defined as the time from first dose until the date of objective progression, or death from any cause, whichever occurs first.
Time Frame: Up to 35 months
Population: The study was terminated during Phase 1 due to strategic reasons; data were not collected or analyzed for this outcome measure in Phase 2.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- IMCnyeso 30-100-300 mcg: IMCnyeso administered intravenously on Days 1, 8, 15, and 22 of each 4-week cycle using an intrapatient escalation regimen (30 mcg on Cycle 1 Day 1, then 100 mcg on Cycle 1 Day 8, then 300 mcg starting on Cycle 1 Day 15)
Arm/Group | Phase 1: IMCnyeso 3 mcg | Phase 1: IMCnyeso 10 mcg | Phase 1: IMCnyeso 30 mcg | Phase 1: IMCnyeso 100 mcg | Phase 1: IMCnyeso 30-100 mcg | Phase 1: IMCnyeso 30-100-180 mcg | IMCnyeso 30-100-300 mcg | Phase 2: Dose Expansion
Number analyzed (Participants) | 4 | 3 | 5 | 3 | 5 | 4 | 5 | 0
Months | 1.8 [0.7 to 2.4] | 1.6 [1.2 to 2.1] | 2.1 [1.9 to 7.8] | 1.9 [1.3 to 1.9] | 2.1 [0.8 to 3.8] | 1.8 [0.9 to 2.1] | 1.4 [1.0 to NA] — Not estimable due to insufficient number of events |

9. Secondary Outcome: Phase 1 and Phase 2: Duration of Response
Description: Duration of response is defined as the time from the date of first documented objective response (CR or PR) until the date of documented disease progression or death.
Time Frame: Up to 35 months
Population: The study was terminated during Phase 1 due to strategic reasons; analysis of duration of response was not able to be performed in Phase 1 because no complete or partial responses were observed and no data were collected for Phase 2.
Arm/Group | Phase 1: Dose Escalation | Phase 2: Dose Expansion
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Phase 1 and Phase 2: Overall Survival
Description: Overall Survival is defined as the time (in months) from the date of randomization to the date of death due to any cause.
Time Frame: Up to 35 months
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 1: IMCnyeso 3 mcg | Phase 1: IMCnyeso 10 mcg | Phase 1: IMCnyeso 30 mcg | Phase 1: IMCnyeso 100 mcg | Phase 1: IMCnyeso 30-100 mcg | Phase 1: IMCnyeso 30-100-180 mcg | Phase 1: IMCnyeso 30-100-300 mcg | Phase 2: Dose Expansion
Number analyzed (Participants) | 4 | 3 | 5 | 3 | 5 | 4 | 5 | 0
Months | 3.3 [2.1 to 5.9] | NA [2.2 to NA] — Not estimable due to insufficient number of events | NA [3.7 to NA] — Not estimable due to insufficient number of events | 9.7 [2.3 to NA] — Not estimable due to insufficient number of events | NA [5.2 to NA] — Not estimable due to insufficient number of events | 7.5 [0.9 to 11.7] | NA [3.7 to NA] — Not estimable due to insufficient number of events |

11. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Time of Last Measurable Concentration (AUC0-last)
Time Frame: Predose and 1, 2, 4, 6, 8, and 12 hours post dose on Cycle 1 Day 1 and Cycle 1 Day 15
Population: The pharmacokinetic analysis set includes participants in the safety analysis set with at least 1 post-dose sample providing evaluable data.
Measure: Mean (Standard Deviation); unit: hr*pg/mL
Arm/Group | Phase 1: IMCnyeso 3 mcg | Phase 1: IMCnyeso 10 mcg | Phase 1: IMCnyeso 30 mcg | Phase 1: IMCnyeso 100 mcg | Phase 1: IMCnyeso 30-100 mcg | Phase 1: IMCnyeso 30-100-180 mcg | Phase 1: IMCnyeso 30-100-300 mcg
Number analyzed (Participants) | 4 | 3 | 4 | 3 | 5 | 4 | 4
hr*pg/mL
  Cycle 1 Day 1: number analyzed (Participants) | 4 | 3 | 4 | 3 | 3 | 4 | 4
  Cycle 1 Day 1 | 12500 (6910) | 17700 (14400) | 132000 (44600) | 295000 (72400) | 182000 (180000) | 78800 (32500) | 127000 (53700)
  Cycle 1 Day 15: number analyzed (Participants) | 4 | 3 | 4 | 2 | 5 | 4 | 1
  Cycle 1 Day 15 | 7270 (4530) | 29500 (35900) | 149000 (70500) | 301000 (223000) | 497000 (260000) | 611000 (330000) | 142000 (NA) — Insufficient number of participants with evaluable data

12. Secondary Outcome: Maximum Observed Plasma Drug Concentration After Single Dose Administration (Cmax)
Time Frame: Predose and 1, 2, 4, 6, 8, and 12 hours post dose on Cycle 1 Day 1 and Cycle 1 Day 15
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Phase 1: IMCnyeso 3 mcg | Phase 1: IMCnyeso 10 mcg | Phase 1: IMCnyeso 30 mcg | Phase 1: IMCnyeso 100 mcg | Phase 1: IMCnyeso 30-100 mcg | Phase 1: IMCnyeso 30-100-180 mcg | Phase 1: IMCnyeso 30-100-300 mcg
Number analyzed (Participants) | 4 | 3 | 4 | 3 | 5 | 4 | 4
pg/mL
  Cycle 1 Day 1: number analyzed (Participants) | 4 | 3 | 4 | 3 | 3 | 4 | 4
  Cycle 1 Day 1 | 1130 (674) | 1530 (1160) | 6850 (1110) | 16100 (961) | 6810 (5290) | 3890 (932) | 6710 (1380)
  Cycle 1 Day 15: number analyzed (Participants) | 4 | 3 | 4 | 2 | 5 | 4 | 1
  Cycle 1 Day 15 | 1090 (634) | 1800 (1290) | 6220 (1450) | 17900 (1910) | 19900 (3570) | 26900 (3930) | 65800 (NA) — Insufficient number of participants with evaluable data

13. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax)
Time Frame: Predose and 1, 2, 4, 6, 8, and 12 hours post dose on Cycle 1 Day 1 and Cycle 1 Day 15
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Phase 1: IMCnyeso 3 mcg | Phase 1: IMCnyeso 10 mcg | Phase 1: IMCnyeso 30 mcg | Phase 1: IMCnyeso 100 mcg | Phase 1: IMCnyeso 30-100 mcg | Phase 1: IMCnyeso 30-100-180 mcg | Phase 1: IMCnyeso 30-100-300 mcg
Number analyzed (Participants) | 4 | 3 | 4 | 3 | 5 | 4 | 4
Hours
  Cycle 1 Day 1: number analyzed (Participants) | 4 | 3 | 4 | 3 | 3 | 4 | 4
  Cycle 1 Day 1 | 1.00 (0.00) | 1.00 (0.00) | 1.00 (0.00) | 1.67 (1.15) | 1.00 (0.00) | 1.25 (0.50) | 1.00 (0.00)
  Cycle 1 Day 15: number analyzed (Participants) | 4 | 3 | 4 | 2 | 5 | 4 | 1
  Cycle 1 Day 15 | 1.00 (0.00) | 1.00 (0.00) | 1.00 (0.00) | 1.00 (0.00) | 1.00 (0.00) | 1.00 (0.00) | 2.00 (NA) — Insufficient number of participants with evaluable data

14. Secondary Outcome: Number of Participants With Anti-IMCnyeso Antibody Formation
Description: Number of participants with positive treatment-boosted or treatment-induced anti-IMCnyeso antibody titers
Time Frame: Up to 35 months
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: IMCnyeso 3 mcg | Phase 1: IMCnyeso 10 mcg | Phase 1: IMCnyeso 30 mcg | Phase 1: IMCnyeso 100 mcg | Phase 1: IMCnyeso 30-100 mcg | Phase 1: IMCnyeso 30-100-180 mcg | Phase 1: IMCnyeso 30-100-300 mcg
Number analyzed (Participants) | 4 | 3 | 5 | 3 | 5 | 4 | 5
Participants | 0 | 0 | 0 | 1 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Up to 35 months
Description: The Safety Analysis Set includes all participants who received at least 1 full or partial dose of study drug in Phase 1; the Phase 2 arm was not started and no data were collected. One participant was sequentially enrolled in two cohorts (10 mcg and 30-100 mcg). Events in either cohort are counted once in the total cohort.
Arm/Group | Phase 1: IMCnyeso 3 mcg | Phase 1: IMCnyeso 10 mcg | Phase 1: IMCnyeso 30 mcg | Phase 1: IMCnyeso 100 mcg | Phase 1: IMCnyeso 30-100 mcg | Phase 1: IMCnyeso 30-100-180 mcg | Phase 1: IMCnyeso 30-100-300 mcg
All-Cause Mortality (participants affected / at risk) | 4/4 | 1/3 | 2/5 | 2/3 | 2/5 | 4/4 | 1/5
Serious Adverse Events (participants affected / at risk) | 3/4 | 1/3 | 1/5 | 1/3 | 2/5 | 3/4 | 3/5
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 5/5 | 3/3 | 5/5 | 4/4 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: IMCnyeso 3 mcg (N=4) | Phase 1: IMCnyeso 10 mcg (N=3) | Phase 1: IMCnyeso 30 mcg (N=5) | Phase 1: IMCnyeso 100 mcg (N=3) | Phase 1: IMCnyeso 30-100 mcg (N=5) | Phase 1: IMCnyeso 30-100-180 mcg (N=4) | Phase 1: IMCnyeso 30-100-300 mcg (N=5)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Muscular haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: IMCnyeso 3 mcg (N=4) | Phase 1: IMCnyeso 10 mcg (N=3) | Phase 1: IMCnyeso 30 mcg (N=5) | Phase 1: IMCnyeso 100 mcg (N=3) | Phase 1: IMCnyeso 30-100 mcg (N=5) | Phase 1: IMCnyeso 30-100-180 mcg (N=4) | Phase 1: IMCnyeso 30-100-300 mcg (N=5)
Anaemia (Blood and lymphatic system disorders) | 4 (7) | 1 (6) | 1 (8) | 0 (0) | 0 (0) | 0 (0) | 2 (8)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (6) | 2 (4) | 2 (2) | 1 (2) | 2 (2) | 2 (4)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (2) | 0 (0) | 1 (1) | 3 (4) | 2 (2) | 1 (4)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (5) | 2 (3) | 4 (11) | 3 (7) | 5 (10) | 3 (8) | 5 (16)
Chills (General disorders) | 0 (0) | 1 (1) | 3 (5) | 2 (7) | 2 (9) | 3 (10) | 3 (14)
Fatigue (General disorders) | 2 (4) | 2 (3) | 2 (2) | 2 (4) | 0 (0) | 2 (4) | 3 (4)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Local swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (4) | 3 (6) | 5 (14)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Corona virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (6)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oxygen saturation decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Breath sounds abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (3) | 3 (6) | 4 (8) | 3 (7) | 2 (4) | 1 (1) | 4 (5)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Phantom pain (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombosis in device (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 3 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 2 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pruritis generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (5) | 1 (1) | 3 (9)
Hypertension (Vascular disorders) | 1 (11) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-02-24): https://cdn.clinicaltrials.gov/large-docs/51/NCT03515551/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-08): https://cdn.clinicaltrials.gov/large-docs/51/NCT03515551/SAP_001.pdf